CLINICAL TRIAL: NCT04746872
Title: Alinity m HR HPV Specimen Collection Study From Women Undergoing Routine Cervical Cancer Screening
Status: Completed | Type: Observational
Sponsor: Abbott Molecular (Industry)
Responsible Party: Sponsor
Other Study IDs: V560-02-20S07-01
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Human Papillomavirus
Keywords: HPV; Virus; Cervical; Cancer; Oncology; Screening; tissue collection; biopsy
MeSH Terms: conditions — Virus Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Alinity m HR HPV: The Alinity m HR HPV IUO assay is a qualitative in vitro test that amplifies and detects HR HPV DNA in cervical cells collected in liquid media. The assay can differentiate between HPV 16, HPV 18, HPV 45 and non-HPV 16/18/45 genotypes [(31/ 33/ 52/ 58) and (35/ 39/ 51/ 56/ 59/ 66/ 68)].
  Interventions: Diagnostic Test: Alinity m HR HPV

INTERVENTIONS:
Diagnostic Test: Alinity m HR HPV — A qualitative in vitro test that amplifies and detects HR HPV DNA in cervical tissue samples.

SUMMARY:
A prospective multicenter interventional study will be conducted to enroll women undergoing routine cervical cancer screening to collect cervical liquid-based cytology (LBC) specimen(s). For all subjects, two cervical specimens will be collected, and one placed into Hologic ThinPrep Pap Test collection kit with PreservCyt Solution (also referred to as ThinPrep specimen) and the other into BD SurePath liquid-based Pap test (also referred to as SurePath specimen). Cytology and HR HPV results will be generated and utilized to determine need for subject referral to colposcopy. Collection of an endocervical curettage (ECC) specimen, and biopsy(ies) if applicable, from women who are referred to colposcopy as a follow up will be conducted according to a standardized protocol. Disease status for each subject will be determined based on cytology, HPV test results, and/or consensus histology review of cervical biopsy specimens.

ELIGIBILITY:
Inclusion Criteria:

Women is eligible if she meets the following:

* Is 25 years of age or older
* Is attending a participating clinic for routine cervical cancer screening following screening guidelines
* Has an intact cervix
* Is willing and able to provide documented informed consent
* Is willing and able to undergo colposcopy, biopsy, and endocervical curettage (ECC) within 12 weeks (≤ 84 days) from the baseline visit, if required
* Is willing and able to allow collection of two cervical cytology specimens

Exclusion Criteria:

A women is ineligible for the study if she meets any of the following criteria:

* Is pregnant at the time of visit or plans to become pregnant within the following 12 weeks
* Has any known medical condition that, in the opinion of the investigator, would result in increased risk of bleeding at biopsy
* Has a known history of excisional or ablative therapy (e.g., LEEP, cone biopsy, cervical laser surgery, or cryotherapy) to the cervix in the last 12 months prior to the baseline visit
* Had a cervical cytology specimen collected within the last 4 months
* Is currently participating in any diagnostic trial for cervical cancer
* Had a complete or partial hysterectomy, either supra cervical or involving removal of the cervix
* Is currently participating or planning to participate in any clinical trial for HPV treatment (for the duration of this study)
* Previous participation in this study

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The participant must be biologically female.
Study Population: Woman who are ≥25 years of age who are high risk humpapillomarius (HPV).
Sampling Method: Non-Probability Sample
Enrollment: 14935 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Disease Progression greater than or equal to (cervical intraepithelial neoplasia) CIN3 | Baseline to 12 weeks
  Diagnosis of greater than or equal to CIN3 (cervical intraepithelial neoplasia) is based on central pathology review panel histologic result.

SECONDARY OUTCOMES:
Disease progression greater than or equal to cervical intraepithelial neoplasia (CIN2) | Baseline to 12 weeks
  Diagnosis of greater than or equal to CIN2 (cervical intraepithelial neoplasia) is based on central pathology review panel histologic result.

CONTACTS AND LOCATIONS:
Locations (62):
- United States (62):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - MedPharmics, LLC, Phoenix, Arizona
  - Desert Bloom Family Medicine / West Valley Research Clinic, LLC, Phoenix, Arizona
  - Quality of Life Medical & Research Centers, LLC, Tucson, Arizona
  - Visions Clinical Research, Tucson, Arizona
  - Northern California Research, Sacramento, California
  - Physicians' Research Options, Lakewood, Colorado
  - Planned Parenthood of Southern New England, New Haven, Connecticut
  - David I Lubetkin, MD, LLC, Boca Raton, Florida
  - Health Awareness INC, Jupiter, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Partners in Womens Health of Jupiter, LLC, Jupiter, Florida
  - Altus Research, Lake Worth, Florida
  - South Florida Clinical Research, Margate, Florida
  - South Miami OB-GYN, Associates, LLC, Miami, Florida
  - Health Awareness, Inc., Port Saint Lucie, Florida
  - Physician Care Clinical Research LLC, Sarasota, Florida
  - Joyce R. Miller, MD, LLC dba South Miami Womens Health an Elligo Health Research Site, South Miami, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Soapstone Center For Clinical Research, Decatur, Georgia
  - The Women's Clinic, Boise, Idaho
  - Clinical Research Prime, Idaho Falls, Idaho
  - Leavitt Women's Healthcare, Idaho Falls, Idaho
  - Providea Health Partners, LLC an Elligo Health Research Site, Mokena, Illinois
  - Women's Health Advantage, Fort Wayne, Indiana
  - Clinical Trials Management, LLC, Covington, Louisiana
  - MedPharmics, LLC, Covington, Louisiana
  - Newman Comprehensive Obgyn, Covington, Louisiana
  - MedPharmics, LLC, Metairie, Louisiana
  - NECCR Fall River LLC, Fall River, Massachusetts
  - Valley Ob-Gyn Clinic, PC and Elligo Health Research Site, Saginaw, Michigan
  - Saginaw Valley Medical Research Group, Saginaw, Michigan
  - Planned Parenthood MN-ND-SD, Saint Paul, Minnesota
  - MedPharmics, Gulfport, Mississippi
  - Meridian Clinical Research, Hastings, Nebraska
  - Women's Clinic of Lincoln, PC, Lincoln, Nebraska
  - Dr. Nader and Associates, Las Vegas, Nevada
  - Rex Garn Mabey, Las Vegas, Nevada
  - Capital Health - Lawrence Ob-Gyn Associates PC, Lawrenceville, New Jersey
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Unified Women's Clinical Research -Raleigh, Raleigh, North Carolina
  - Unified Women's Clinical Research- Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Cleveland MacDonald Women's Hospital, Cleveland, Ohio
  - Hilltop Obstetrics & Gynecology, Inc., Franklin, Ohio
  - The Ohio State University Obstetrics and Gynecology Worthington, Worthington, Ohio
  - OB GYN Associates of Erie, Erie, Pennsylvania
  - VitaLink Research - Greenville, Greenville, South Carolina
  - Tribe Clinical Research dba Mountain View Clinical Research, Greer, South Carolina
  - Medical Research Center of Memphis, LLC, Memphis, Tennessee
  - Women's Health Texas, LLC (Elligo), Austin, Texas
  - Hill Country OB/GYN Associates, Austin, Texas
  - Austin Area Obgyn, PLLC, Austin, Texas
  - Christina Sebestyen MD, P.A. dba OBGYN North, Austin, Texas
  - Nueces County Women's Clinic dba Corpus Christi Women's Clinic an Elligo Health Research Site, Corpus Christi, Texas
  - Advanced Research Associates, Corpus Christi, Texas
  - Ventavia Research Group, Fort Worth, Texas
  - TMC Life Research, Inc., Houston, Texas
  - Cedar Health Research, LLC_Avacare West, Irving, Texas
  - Medical Colleagues of Texas, LLP, Katy, Texas
  - Physicians Research Options, Draper, Utah
  - Tidewater Clinical Research Inc, Norfolk, Virginia